CLINICAL TRIAL: NCT06276335
Title: Influence of Timing of Implant Placement on Early Healing Molecular Events: A Two-centre, Parallel Group, Pilot Study
Brief Title: Influence of Timing of Implant Placement on Early Healing Molecular Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRAS:322440
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant; Healing Wound; Biomarkers; Saliva
Keywords: Implant placement protocol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant placement and conventional loading (Test) (Experimental): In this group, a dental implant will be placed on the same day as tooth extraction and loaded after 3 months
  Interventions: Other: Immediate implant placement and guided bone regeneration (Test)
- Late implant placement and conventional loading (Control) (Active Comparator): In this group, a dental implant will be placed after complete bone healing (4 - 6 months after tooth extraction) and loaded after 3 months
  Interventions: Other: Late implant placement and guided bone regeneration (Control)

INTERVENTIONS:
Other: Immediate implant placement and guided bone regeneration (Test) — In this group, immediately after tooth extraction, a tapered bone level implant (Straumann BLX Implant System, Roxolid, Straumann AG, Basel, Switzerland) will be placed in an ideal prosthetically oriented position to achieve primary stability following the manufacture's guidelines. A prefabricated surgical template based on 3D pre-extraction planning will be used to place the implant. The jumping distance between the implant and the residual buccal bone will be measured and filled with slow resorption bone graft material (Bio-Oss®, Geistlich, Wolhusen, Switzerland) as per standard of practice.
  Arms: Immediate implant placement and conventional loading (Test)
Other: Late implant placement and guided bone regeneration (Control) — A tapered bone level implant (Straumann BLX Implant System, Roxolid, Straumann AG, Basel, Switzerland) will be placed after complete bone healing (4 - 6 months after tooth extraction) in an ideal prosthetically oriented position to achieve primary stability following the manufacture's guidelines. Guided bone regeneration (GBR) will be performed simultaneously with the aim to re-establish the bone contour and treat any fenestration/dehiscence if needed. A bovine osteoconductive graft (Bio-Oss®, Geistlich, Wolhusen, Switzerland) will be loosely compacted on the buccal aspect of the implant and covered with a collagen membrane (Bio-Gide®, Geistlich, Wolhusen, Switzerland).
  Arms: Late implant placement and conventional loading (Control)

SUMMARY:
Dental implants have been on the market for several years and they are routinely used to replace single/multiple missing teeth with a high success rate. However, there is still a limited number of studies comparing the influence of timing of implant placement on wound healing. In addition, there is no data available on the signaling pathways and the expression of healing biomarkers involved in the early stages of osseointegration after immediate implant placement (IP) or delayed implant placement (DP).

The primary objective of this study is to describe changes in the expression of inflammatory, angiogenesis and osseous biomarkers of saliva at 1, 3, 7, 15 and 30 days and of PICF at 3, 7, 15 and 30 days after immediate implant placement (IP) compared with delayed placement (DP).

DETAILED DESCRIPTION:
This is a two-centre prospective, parallel-group pilot study which will consist of 10 to 11 visits over a minimum period of 16 months. The study will take place at the Centre for Oral Clinical Research (COCR), at the Institute of Dentistry, Barts and The London School of Medicine and Dentistry, Queen Mary University of London (main centre), United Kingdom and at the Implant Research Centre, School of Dental Medicine, University of Belgrade, in accordance with local guidelines and procedures/ interventions detailed below.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥25 years old
* Good/controlled medical and psychological health
* Good oral hygiene (FMPS≤20%)
* Presence of a tooth in the aesthetic region (from incisor to second premolar) in need of extraction and further oral rehabilitation with a single dental implant.
* For the IP group, the extraction socket should fulfil the following parameters, as described by the 5th ITI consensus [46]: intact socket wall; facial bone wall ≥1mm in thickness; no acute infection at the site; availability of bone apical and palatal to the socket to provide primary stability.
* At least one neighbouring natural tooth.
* A functional occlusion with a minimum of four occlusal units (i.e., pairs of occluding posterior teeth).
* Willingness to read and sign a copy of the Informed Consent Form (ICF) after reading the Patient Information Sheet (PIS), and after the nature of the study has been fully explained and potential questions fully answered.

Exclusion Criteria:

* Any known systemic disease severely affecting bone metabolism (e.g., Cushing's syndrome, Crohn's disease, rheumatoid arthritis, osteoporosis or diabetes type I and uncontrolled diabetes type II).
* Self-reported HIV or viral hepatitis.
* Self-reported alcoholism or chronic drug abuse.
* Smokers (including current smokers or former smokers who had quit for < 3 months); patients reporting use of vape/e-cigarettes will also be excluded.
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing, which can affect interpretation of study results).
* Chronic treatment (i.e., 2 weeks or more) with any medication known to affect oral status or bone metabolism (e.g., bisphosphonates, hormone replacement therapy, immunosuppressants) within 1 month before baseline visit.
* Chronic treatment with anticoagulants (including Aspirin), corticosteroids, immunosuppressants or other medications that may influence blood coagulation/count.
* Antibiotic or anti-inflammatory therapy during the month preceding the baseline exam.
* Untreated caries lesions and untreated/uncontrolled periodontal disease; If patients require periodontal treatment (non-surgical and/or surgical), this will be arranged outside the study protocol and completed prior to enrolment;
* Inadequate keratinized tissue width (<2 mm) in the mid-buccal aspect of the area to be treated in the study.
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene in the area of implant placement.
* Patients requiring maxillary sinus lift surgery before implant placement.
* Self-reported bruxism.
* Patients not willing to receive animal-derived biomaterials for GBR.
* Patients suffering from a known psychological disorder or with limited mental capacity or language skills such that study information could not be understood, informed consent could not be obtained, or simple instructions could not be followed.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the expression of inflammatory, angiogenesis and osseous biomarkers of PICF and saliva | 1, 3, 7, 15 and 30 days after immediate or delayed implant placement
  The expression of inflammatory, angiogenesis and osseous biomarkers of PICF at 3, 7, 15 and 30 days after immediate implant placement (IP) or delayed placement (DP) and of saliva at day 1, 3, 7, 15 and 30

SECONDARY OUTCOMES:
Blood flow changes | immediately after, 1, 3, 7, 15 and 30 days after immediate or delayed implant placement
  Blood flow changes immediately after, at 1, 3, 7, 15 and 30 days after implant placement
Soft tissue volume changes | immediately after,1, 3, 7, 15, 30 days and 3 months after immediate or delayed implant placement, at loading and 6 months after implant loading
  Soft tissue volume changes immediately after, at 1, 3, 7, 15, 30 days and 3 months after immediate or delayed implant placement, at loading and 6 months after implant loading
Peri-implant bone level | 6 months after implant loading
  Peri-implant bone level 6 months after loading, using CBCT images
Full mouth plaque score (FMPS) | 6 months after implant loading
  FMPS will be recorded as a percentage of total surfaces (6 sites per tooth/implant), which reveal the presence of plaque. A binary score will be assigned to each surface (1 for plaque present, 0 for absent).
Full mouth bleeding score (FMBS) | 6 months after implant loading
  FMBS will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of bleeding within 10 - 30 seconds following periodontal probing. A binary score will be assigned to each surface (1 for bleeding present, 0 for bleeding absent).
Probing pocket depth (PPD) | 6 months after implant loading
  PPD will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/ implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual).
Gingival recession (REC) | 6 months after implant loading
  REC will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/ implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual).
Clinical attachment level (CAL) | 6 months after implant loading
  CAL will be calculated considering the values for PPD and REC in mm
Suppuration | 6 months after implant loading
  Suppuration will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of suppuration following periodontal probing. A binary score will be assigned to each surface (1 for suppuration present, 0 for suppuration absent).
Patient satisfaction at 6 months after loading | 6 months after implant loading
  Patient satisfaction regarding the overall implant treatment using a subjective outcome questionnaire at 6 months post loading.
Changes in the pink esthetic score (PES) | 6 months after implant loading
  Changes in the pink esthetic score (PES) from loading to 6 months after loading
Changes in the white esthetic score (WES) | 6 months after implant loading
  Changes in the white esthetic score (WES) from loading to 6 months after loading
Changes in the papilla fill index (PFI) | 6 months after implant loading
  Changes in the papilla fill index (PFI) from loading to 6 months after loading
Implant survival | 6 months after implant loading
  Implant functionally present in the mouth

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, Principal Investigator — QMUL
Locations (1):
- Centre for Oral Clinical Research, London, United Kingdom